CLINICAL TRIAL: NCT06034327
Title: Efficacy in Controlling Myopia in Young Children Using a Novel Spectacle Lens
Acronym: EUCALYPTUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SightGlass Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPRO-2304-001
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Myopia; Juvenile Myopia; Myopia Progression
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and parents of participants will be masked. Investigational site staff tasked with measuring key primary variables will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Test Arm 1 (Experimental): Single vision, impact-resistant spectacle lenses
  Interventions: Device: Single vision, impact-resistant spectacle lenses; Test Arm
- Test Arm 2 (Other): Single vision, impact-resistant spectacle lenses
  Interventions: Device: Single vision, impact-resistant spectacle lenses; Control Arm

INTERVENTIONS:
Device: Single vision, impact-resistant spectacle lenses; Test Arm — Use of single vision, impact-resistant spectacle lenses may reduce the rate of progression of juvenile myopia
  Arms: Test Arm 1
Device: Single vision, impact-resistant spectacle lenses; Control Arm — Single vision, impact-resistant spectacle lenses
  Arms: Test Arm 2

SUMMARY:
This is a conventional efficacy trial to validate the results from previous clinical trials for younger children; the 12-month efficacy results will be used to predict the 3-year treatment efficacy.

This is a randomized, controlled (1:1), multisite, subject- and observer-masked, 2-arm parallel group study.

ELIGIBILITY:
Inclusion Criteria:

1. Children 6 - 8 years of age (inclusive) at time of informed consent/assent;
2. Spherical equivalent refractive error between -0.75 and -4.50 D inclusive (by manifest refraction) in each eye;
3. Astigmatism if present, less than or equal to -1.25 DC (by manifest refraction) in each eye;
4. Best corrected visual acuity by manifest refraction of +0.10 logMAR (20/25 Snellen equivalent) or better in each eye;
5. The difference in spherical equivalent power between the two eyes (anisometropia based on manifest refraction) must be less than or equal to 1.50 D;
6. Agree to wear the assigned spectacles constantly except for sleeping, swimming, or other activities in which spectacle wear would be dangerous or otherwise not possible (minimum of 10 hours per day);
7. Ability to comply with study procedures, including high and low contrast visual acuity, axial length, and cycloplegic autorefraction measurements taken for both eyes at the baseline visit;
8. Willingness to participate in the trial for 24 months without contact lens wear;
9. The subject's parent(s) or legal guardian(s) must read, understand and sign the Statement of Informed Consent and receive a fully executed copy of the form.

Exclusion Criteria:

1. Subject has previously or currently wears contact lenses (greater than 1-month usage);
2. Current or prior use of bifocals, progressive addition spectacle lenses
3. Current or prior use of any myopia control treatment (e.g., atropine, multifocal contact lenses, orthokeratology);
4. Amblyopia in either eye;
5. Strabismus by cover test at far (4 m) or near (40 cm) wearing distance correction;
6. Any ocular or systemic conditions that could influence refractive development or status [e.g., keratoconus, congenital glaucoma, ocular trauma, diabetes, Marfan syndrome or other connective tissue disorder, Down's syndrome, family history of poor night vision (to prevent against enrolling subjects with congenital stationary night blindness)];
7. Known allergy to proparacaine, tetracaine, or tropicamide;
8. Participation in any investigational clinical study within 30 days of the Baseline visit;
9. Subject's sibling or other household member is already enrolled in this trial.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Spherical equivalent refraction | 12 months
  Change in spherical equivalent refraction from baseline

SECONDARY OUTCOMES:
Axial length | 12 months
  Change in axial length from baseline

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Elsa Pao, OD, Oakland, California
  - Scripps Poway Eyecare, San Diego, California
  - Pacific Rims Optometry, San Francisco, California
  - Paje Optometric, Santa Ana, California
  - Omega Vision Center, Longwood, Florida
  - Marietta Eye Clinic, Marietta, Georgia
  - Ilinois College of Optometry, Chicago, Illinois
  - Kannarr Eye Care, Pittsburg, Kansas
  - New England College of Optometry, Boston, Massachusetts
  - Advanced Eyecare PC, Raytown, Missouri
  - Athens Eye Care, Athens, Ohio
  - Procare Vision Centers, Inc., Granville, Ohio
  - Texas State Optical - Dowlen, Beaumont, Texas
  - Bellaire Family Eye Care, Bellaire, Texas